CLINICAL TRIAL: NCT01018290
Title: Preoperative Non-Invasive Motor Mapping in Tumor Surgery by Navigated Transcranial Magnetic Stimulation
Brief Title: Navigated Transcranial Magnetic Stimulation in Tumor Surgery
Status: Terminated | Type: Observational
Why Stopped: Recruitment goals not met
Sponsor: Nexstim Ltd (Industry)
Responsible Party: Alexandra Golby, MD, Neurosurgery, Brigham and Women's Hospital, Partners Healthcare System, Harvard Medical School
Other Study IDs: 2008-P-002325/2
Record Dates: First submitted 2009-11-20; First posted 2009-11-23 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2011-06

CONDITIONS: Brain Tumors
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Navigated TMS examination: 20 patients with brain tumor in the vicinity of the central motor region scheduled for elective surgery will undergo pre-operative Navigated TMS examination to determine the localization of primary motor cortex and motor representation areas of specific muscles

SUMMARY:
Maximizing surgical removal of brain tumors while minimizing neurologic deficits is challenging. Functional brain tissue may reside close to or even within the abnormality, and inadvertent removal or disturbance of such areas can result in neurologic deficits. At present, the gold standard for identifying critical motor areas in tumor surgery is intraoperative invasive direct current stimulation (DCS) through a handpiece. More recently, new non-invasive preoperative method for brain mapping, functional magnetic resonance imaging (fMRI), may be used to identify the eloquent motor areas. fMRI signals used in localization of the motor areas are generated when the brain is activated during the performance of specific motor tasks. However, as fMRI signals are also generated by sensory input, the resulting fMRI map may include sensory as well as motor areas.

Nexstim has developed a Navigated Brain Stimulation (NBS) system that uses TMS with a software based Navigational System that together may have more specific spatial accuracy.

This study aims to determine whether navigated TMS is able to identify the eloquent motor cortical areas in patients with brain tumors and to determine the clinical accuracy of the procedure by comparing it to results obtained by intraoperative DCS and fMRI.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects 18 years of age and over.
* A brain tumor in the vicinity of the central region.
* Mild (BMRC grade 4/5) or no paresis.
* Obscured anatomy of the central region due to the mass effect/infiltrating growth pattern of the lesion
* Scheduled for elective surgery under general or local anesthesia.
* No other known brain abnormalities by history or by structural MRI.
* Mentally and physically able to undergo MR imaging (fMRI, DTI) and navigated TMS studies
* Signed informed consent form.

Exclusion Criteria:

* Implanted metallic parts of implanted electronic devices, including pacemakers, defibrillators, or implant medication pump.
* Pregnant or trying to become pregnant.
* History of alcohol abuse, illicit drug use or drug abuse or significant mental illness
* Hypertensive or hypotensive condition.
* Any condition that would prevent the subject from giving voluntary informed consent.
* An implanted brain stimulator.
* Aneurysm clip or other metal in the head (except mouth
* Enrolled or plans to enroll in an interventional trial during this study.
* Scalp wounds or infections.
* Claustrophobia precluding MRI
* Frequent seizures (>1/week)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 20 patients with brain tumor in the vicinity of the central motor region scheduled for elective surgery.Patients aged 18 and over with no other brain abnormalities.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2009-11; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Distance between motor representation area localization by NBS to that determined by DCS | immediate post-operative period
Comparison of DTI results based on using NBS motor representations as seed to those obtained using DCS results as seeds | immediate post-operative period

SECONDARY OUTCOMES:
Comparison of the relative distance of NBS anf fMRI identified motor representations to those determined by DCS | immediate post-operative period
Assess safety of navigated TMS in this patient population by capturing all Serious Adverse Events | During and after navigated TMS examination

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Golby, MD, Principal Investigator — Brigham and Women's Hospital Harvard Medical School
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States